CLINICAL TRIAL: NCT05566899
Title: Primary Objective: The Primary Objective of the Study is to Evaluate the Acceptability and Feasibility of EGD-SC
Brief Title: Pilot Study of Stomach Cancer Early Detection and Prevention With Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Haejin In, Surgical Oncology Associate Professor of Surgery, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 072211; Pro2022001252 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-07-05; First posted 2022-10-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer
Keywords: H.pylori infection; chronic atrophic gastritis
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: A single-center, open label pilot study that will evaluate the acceptability and feasibility of EGD at time of routine screening colonoscopy (EGD-SC). The Pre-Study Screening is day -30 to day 0; EDG at time of routine screening colonoscopy and follow-up day five to seven.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- EGD at time of routine screening colonoscopy (Experimental): This happens on Day 0. Screening for EGD, biopsy samples from esophagus, stomach, gastrointestinal junction, and duodenum AE's.
  Interventions: Procedure: esophagogastroduodenoscopy (EGD)

INTERVENTIONS:
Procedure: esophagogastroduodenoscopy (EGD) — After colonoscopy, the patient will undergo the EGD at which time biopsy specimens will be obtained.
  Participants will also be provided with a home stool collection kit which they can bring to the endoscopy visit or mail back. Satisfaction questions will be administered 3-7 days after EGD-SC

SUMMARY:
Screening esophagogastroduodenoscopy (EGD )provides three distinct opportunities to decrease gastric cancer (GC) morbidity and mortality. has potential to discover cancer in early stages before the onset of symptoms, leading to higher rates of survival. Second, premalignant lesions such as adenomatous polyps, intestinal metaplasia and dysplasia can be discovered and removed with local resection, akin to polypectomies during screening colonoscopies, preventing the development of cancer. Third, EGD discovery and treatment of active Helicobacter pylori (HP) infection of the stomach provides an opportunity for primary prevention of GC.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the acceptability and feasibility of EGD-SC.

The secondary objectives are:

1. Estimate Median added time needed for EGD at the time of routine screening colonoscopy
2. Estimate the frequencies of adverse events
3. Estimate the percentage of pre-cancer and cancerous lesions including H. pylori infection, chronic atrophic gastritis, IM, dysplasia and GC among this high GC risk population
4. Investigate whether high-risk racial/ethnicity groups have different likelihood of uptake of EGD, and whether the likelihood is associated with patient beliefs, attitudes and knowledge of GC, perceptions of risk, motivators and barriers, and sociocultural factors, as well as patient preference and satisfaction with EGD-SC

ELIGIBILITY:
Inclusion Criteria:

* Have provided signed informed consent for the trial
* Aged =40 and =80 years at the time of informed consent
* Not planned to undergo EGD and not had EGD in the last five years
* Planned to undergo colonoscopy
* Half of the recruited subjects will be from high-risk groups
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Persons with total gastrectomy
* Persons with anatomic alteration that precludes EGD
* Medical conditions that substantially increase risks for EGD
* Had EGD in the last five years

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability and feasibility of EGD-SC measured by Linear Scale | Pre-Study Screening Day -30 to day0
  To achieve the goal of assessing feasibility of EDG-SC as well as estimates of effect size needed to determine sample size and power for the planned study, the investigator will collect data on the number of participants contacted, number eligible, and number who agree to EGD-SC.

SECONDARY OUTCOMES:
Number of participants with AE's will be measured by the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 5.0 | From the time of consent to through five calendar days after screening/treatment
  Adverse events (AEs) will be evaluated and graded using the Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 5.0

OTHER OUTCOMES:
Acceptability and feasibility of EGD-SC measured by Linear Scale | Pre-Study Screening Day -30 to day 0
  Linear Scale eligible for the study. The Wilcoxon signed-rank test will be used to assess the participants responses to EGD.

CONTACTS AND LOCATIONS:
Overall Officials: Haejin In, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No